CLINICAL TRIAL: NCT05350878
Title: Implementing Mobile Technology for Unhealthy Alcohol Use in Emergency Departments
Brief Title: Implementing Mobile Technology for Unhealthy Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Northwell Health (Other); Partnership to End Addiction (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Megan O'Grady, Assistant Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: O22-184-1; R21AA029734 (NIH)
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Drinking
Keywords: Implementation Science; Text Messaging; Unhealthy Alcohol Use; Mobile Health; mHealth
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Parallel Cluster Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implementation Intervention (Experimental): Through virtual and in-person meetings, the internal/external facilitation team will support sites in utilizing the multi-component implementation strategy for 7 months
  Interventions: Other: Implementation Intervention
- Implementation as Usual (No Intervention): In control 'implementation as usual' sites, no facilitation or implementation strategies will be provided. Controls will receive 1) an informational session on the text intervention during grand rounds/staff meetings and 2) flyers to provide patients with intervention enrollment information.

INTERVENTIONS:
Other: Implementation Intervention — Virtual and in-person implementation support
  Arms: Implementation Intervention

SUMMARY:
Scalable approaches are needed to support patients identified in the emergency department as unhealthy alcohol users and text messaging intervention approaches are a promising solution. However, the process of providers making text messing interventions for unhealthy alcohol use available to patients in an efficient way within already busy and overburdened emergency department workflows (i.e., implementation in real-world emergency department settings) and patients adopting them remains a new area of research. Study investigators will examine barriers and facilitators to the adoption of text messaging interventions for unhealthy alcohol use in emergency departments and use a stakeholder-engaged process to develop and test practical implementation strategies that could provide much needed support to patients who screen positive while reducing burden on emergency departments.

DETAILED DESCRIPTION:
Unhealthy alcohol use (UAU) is one of the leading causes of premature mortality among adults in the United States and has been increasing during the COVID-19 pandemic. UAU is more frequent among emergency department (ED) patients than in the general population and ED visits involving alcohol consumption have increased in recent years. Substance use has been described as the most important modifiable health behavior in the ED, and the ED has been highlighted as a key setting to intervene with UAU individuals. Consequently, health systems across the country need low burden, scalable ways to intervene with individuals but often have limited time and resources. Mobile technologies have been suggested as a solution to assist EDs in addressing UAU and one of the lowest burden, scalable approaches are text messaging interventions. Text messaging interventions for ED and trauma patients and other populations have shown good outcomes, including reductions in drinking quantity and frequency. Despite strong research support and promise for scalability, there is little evidence that technology-based behavioral health interventions can be effectively implemented into healthcare settings. There are few studies in which technology interventions for behavioral health are put into real world healthcare settings; those that have been conducted show that the benefits seen in randomized trials are often not realized. While EDs are promising venues for addressing UAU using text messaging interventions, the process of providers making them available to patients in an efficient way within already busy and overburdened ED workflows (i.e., implementation in real-world ED settings) and patients adopting them remains a new area of research. This proposal builds on the longstanding collaboration of our interdisciplinary team on the implementation of substance use screening and brief interventions in healthcare settings. In response to the NIH Notice of Special Interest for Research in the Emergency Setting, the investigators propose to examine potential barriers and facilitators to staff offering and patients accepting a text messaging intervention in the ED. The investigators will then use a stakeholder-engaged Intervention Mapping process to develop a multi-component implementation strategy for EDs. Finally, the investigators will conduct a mixed method 2-arm cluster-randomized pilot study in 4 EDs that serve ~13,000 UAU patients per year to assess the feasibility, acceptability and preliminary effectiveness of the implementation strategy. The Integrated Promoting Action on Research Implementation in Health Services (i-PARIHS) framework will guide study activities. Low burden technology, like text messaging, along with targeted implementation support and strategies driven by identified barriers and facilitators could sustain large-scale ED-based alcohol screening programs and provide much needed support to patients who screen positive while reducing burden on EDs. The proposed study would be the first to develop and test this targeted implementation strategy. This 2-year R21 will prepare for a future, larger, fully-powered hybrid effectiveness-implementation trial.

ELIGIBILITY:
Patient Inclusion Criteria

* Emergency department patient at one of the participating sites
* 18 years or older
* English-language fluency
* Owing a text-capable phone

Staff Inclusion Criteria:

* Emergency department staff and providers who work in the intervention sites
* Employed full or part time by the participating health system

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Implementation Effectiveness | 5-month intervention period
  The proportion of eligible patients who enroll in the alcohol text messaging intervention

SECONDARY OUTCOMES:
Implementation Feasibility using the Feasibility of Intervention Measure (FIM) | 6-months post-intervention
  Feasibility of text messaging implementation strategy
Implementation Acceptability using the Acceptability of Intervention Measure (AIM) | 6-months post-intervention
  Acceptability of text messaging implementation strategy

CONTACTS AND LOCATIONS:
Overall Officials: Megan A O'Grady, PhD, Principal Investigator — UConn Health
Locations (1):
- Northwell Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared in the NIAAA Data Archive
Time Frame: Data will be available at the end of the study
Access Criteria: Per NIAAA archive access criteria
URL: https://www.niaaa.nih.gov/research/niaaa-data-archive

REFERENCES:
- [Derived] O'Grady MA, Kapoor S, Harrison L, Kwon N, Suleiman AO, Muench FJ. Implementing a text-messaging intervention for unhealthy alcohol use in emergency departments: protocol for implementation strategy development and a pilot cluster randomized implementation trial. Implement Sci Commun. 2022 Aug 6;3(1):86. doi: 10.1186/s43058-022-00333-y. PMID 35933560